CLINICAL TRIAL: NCT00637806
Title: A Randomized, Double-blind, Placebo-controlled Study of Megestrol Acetate Concentrated Suspension for the Treatment of Cancer-associated Anorexia in Subjects With Cancer of Multiple Types
Brief Title: Treatment of Cancer-associated Anorexia Using Megestrol Acetate Concentrated Suspension
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulty finding the required patient population
Sponsor: Par Pharmaceutical, Inc. (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 100.2.C.005 TRANSFERRED
Record Dates: First submitted 2008-03-11; First posted 2008-03-18 (Estimated); Results first posted 2016-05-02 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-03

CONDITIONS: Anorexia; Cachexia; Weight Loss
Keywords: Megestrol acetate; Anorexia; Cachexia; Cancer; Unintended weight loss; Body weight; Appetite; Megace ES
MeSH Terms: conditions — Anorexia; Cachexia; Weight Loss; Neoplasms; Body Weight | interventions — Megestrol Acetate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Megestrol acetate concentrated suspension 110 mg/mL
  Interventions: Drug: Megestrol acetate concentrated suspension 110 mg/mL
- 2 (Active Comparator): Megestrol acetate concentrated suspension 60 mg/mL
  Interventions: Drug: Megestrol acetate concentrated suspension 60 mg/mL
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Megestrol acetate concentrated suspension 110 mg/mL — Megestrol acetate concentrated suspension 110 mg/mL given as an oral dose of 550 mg (5 mL) once per day for 56 days, with an optional 28 days extension phase
  Other Names: Megace ES
  Arms: 1
Drug: Megestrol acetate concentrated suspension 60 mg/mL — Megestrol acetate concentrated suspension 60 mg/mL given as an oral dose of 300 mg (5 mL) once per day for 56 days, with an optional 28 days extension phase
  Other Names: Megace ES
  Arms: 2
Drug: Placebo — Placebo oral suspension, 5 mL once daily
  Arms: 3

SUMMARY:
To compare the effect of megestrol acetate concentrated suspension and placebo on caloric intake in patients with cancer-associated anorexia.

ELIGIBILITY:
Inclusion Criteria:

* Cancer of multiple types in stage II, III, or IV and not a candidate for chemotherapy; but may have been receiving radiation therapy
* Fair, poor, or very poor appetite
* Cancer-associated anorexia/cachexia (documented weight loss of 2% over the prior week, or at least 5% within past 30 days, or at least 7.5% over prior 3 months, or at least 10% over prior 6 months)
* Weight loss perceived to be associated with diminished appetite
* Eastern Cooperative Oncology Group Performance score of 0, 1, or 2
* Life expectancy greater than 3 months
* Alert and mentally competent to complete study assessments
* Women of child-bearing potential required to use an adequate and reliable method of contraception. Post-menopausal women have to have been so for at least 1 year
* Screening laboratory values must not be clinically significant (some exceptions per protocol)

Exclusion Criteria:

* Brain, or head and neck tumors that may interfere with food consumption
* AIDS-related wasting
* Radiation therapy to head and neck, abdomen, or pelvis within past 6 weeks, or for whom radiation therapy is anticipated during the study such that the result may interfere with food consumption
* Presence of conditions that interfere with oral intake or ability to swallow
* Absence of normally functioning gut
* Known mechanical obstruction of the alimentary or biliary tract, or malabsorption syndrome
* Intractable or frequent vomiting
* Clinically significant diarrhea
* History of thromboembolic events, or on long-term anticoagulation for thromboembolism
* Uncontrolled diabetes mellitus, or symptomatic hypoadrenalism
* Poorly controlled hypertension or congestive heart failure
* Pregnant/lactating females, or planning on becoming pregnant
* Use of appetite stimulants within past 30 days
* Use of parenteral nutrition or tube feedings within past 1 week
* Chronic use of steroids within past 3 months (intermittent short-term use allowed)
* Current use of illicit substances
* Allergy, hypersensitivity, or other contraindication to megestrol acetate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2006-06; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn D Kramer, MD, Study Chair — Par Pharmaceutical, Inc.; Janet Bull, MD, Principal Investigator — Four Seasons Hospice and Paliative Care; Veena Charu, MD, Principal Investigator — Pacific Cancer Medical Center, Inc.; Bart Frizzell, MD, Principal Investigator — Wake Forest University, Dept of Radiation Oncology; Mehool Patel, MD, Principal Investigator — Summit Oncology Associates, Inc.
Locations (4):
- United States (4):
  - Pacific Cancer Medical Center, Inc., Anaheim, California
  - Four Seasons Hospice and Paliative Care, Flat Rock, North Carolina
  - Wake Forest University, High Point, North Carolina
  - Summit Oncology Associates, Inc., Akron, Ohio

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After screening, eligible subjects were randomized to treatment in the double-blind phase. After completing the double-blind phase or discontinuing due to specific weight loss criteria, eligible subjects could enter an open-label extension phase.
Groups:
- DB MA-CS 550 mg/Day: Megestrol acetate concentrated suspension (MA-CS; 110 mg/mL) administered orally once every 24 hours (q24h), for a daily dose of 550 mg per day (5 mL dose) in the 8-week double-blind (DB) phase
- DB MA-CS 300 mg/Day: MA-CS (60 mg/mL) administered orally q24h, for a daily dose of 300 mg per day (5 mL dose) in the 8-week DB phase
- DB Placebo: Placebo suspension administered orally q24h (5 mL dose) in the 8-week DB phase
- OL MA-CS 550 mg/Day: MA-CS (110 mg/mL) administered orally q24h, for a daily dose of 550 mg per day (5 mL dose) in the 4-week open-label (OL) extension phase
Period: Double-blind Phase
Arm/Group | DB MA-CS 550 mg/Day | DB MA-CS 300 mg/Day | DB Placebo | OL MA-CS 550 mg/Day
Started | 2 | 0 | 2 | 0
Completed | 0 | 0 | 1 | 0
Not Completed | 2 | 0 | 1 | 0
Not completed — Study Discontinued | 2 | 0 | 1 | 0
Period: Extension Phase
Arm/Group | DB MA-CS 550 mg/Day | DB MA-CS 300 mg/Day | DB Placebo | OL MA-CS 550 mg/Day
Started | 0 | 0 | 0 | 1
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 1
Not completed — Study Discontinued | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All subjects who received at least 1 dose of study medication and who had at least 1 on-therapy safety assessment
Groups:
- DB MA-CS 550 mg/Day: MA-CS (110 mg/mL) administered orally q24h, for a daily dose of 550 mg per day (5 mL dose) in the 8-week DB phase
- Total: Total of all reporting groups
Arm/Group | DB MA-CS 550 mg/Day | DB MA-CS 300 mg/Day | DB Placebo | Total
Number analyzed (Participants) | 2 | 0 | 2 | 4
Age, Categorical [Number; unit: participants]
  <=18 years | 0 |  | 0 | 0
  Between 18 and 65 years | 1 |  | 0 | 1
  >=65 years | 1 |  | 2 | 3
Gender [Number; unit: participants]
  Female | 1 |  | 0 | 1
  Male | 1 |  | 2 | 3
Ethnicity (NIH/OMB) [Number; unit: participants]
  Hispanic or Latino | 0 |  | 0 | 0
  Not Hispanic or Latino | 2 |  | 2 | 4
  Unknown or Not Reported | 0 |  | 0 | 0
Race (NIH/OMB) [Number; unit: participants]
  American Indian or Alaska Native | 0 |  | 0 | 0
  Asian | 0 |  | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 |  | 0 | 0
  Black or African American | 0 |  | 0 | 0
  White | 2 |  | 1 | 3
  More than one race | 0 |  | 0 | 0
  Unknown or Not Reported | 0 |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 |  | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Average Daily Caloric Intake Over the Course of the 8-week Double-blind Phase
Description: The Nutrition Data System for Research (NDSR) was used to determine nutrient and caloric value for foods and beverages consumed and recorded by subjects over a 3-day assessment period prior to each visit. Total number of calories consumed during each 3-day assessment was averaged over available values to determine the week's daily caloric intake value.
Time Frame: 8 weeks
Population: Results not analyzed due to early termination of the study
Arm/Group | DB MA-CS 550 mg/Day | DB MA-CS 300 mg/Day | DB Placebo
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Change in Weight Over the Course of the 8-week Double-blind Phase
Time Frame: Baseline, Week 1, 2, 3, 4, 6, and 8
Population: Results not analyzed due to early termination of the study
Arm/Group | DB MA-CS 550 mg/Day | DB MA-CS 300 mg/Day | DB Placebo
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Changes in Body Composition as Measured by Bioelectric Impedance Analysis (BIA) at Week 4 and Week 8 Relative to Baseline
Time Frame: Baseline, Week 4 and Week 8
Population: Results not analyzed due to early termination of the study
Arm/Group | DB MA-CS 550 mg/Day | DB MA-CS 300 mg/Day | DB Placebo
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Change in Appetite Over the 8-week Double-blind Phase as Measured by a VAS Appetite Scale
Description: Subjects marked 6 items on a visual analog scale (VAS) appetite scale including feeling not hungry to hungry, not nauseated to nauseated, empty to full, not satiated to satiated; weak to strong desire to eat; and ability to eat none to a large amount of food
Time Frame: Baseline, Weeks 1, 2, 3, 4, 6 and 8
Population: Results not analyzed due to early termination of the study
Arm/Group | DB MA-CS 550 mg/Day | DB MA-CS 300 mg/Day | DB Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Approximately 98 days (from informed consent through 7 days following the last dose of study drug or up until the last protocol-specified study visit, whichever occurred later)
Groups:
- OL MA-CS 550 mg/Day: MA-CS (110 mg/mL) administered orally q24h, for a daily dose of 550 mg per day (5 mL dose) in the 4-week OL extension phase
Arm/Group | DB MA-CS 550 mg/Day | DB MA-CS 300 mg/Day | DB Placebo | OL MA-CS 550 mg/Day
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0 | 1/2 | 1/1
Other Adverse Events (participants affected / at risk) | 1/2 | 0/0 | 2/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DB MA-CS 550 mg/Day (N=2) | DB MA-CS 300 mg/Day (N=0) | DB Placebo (N=2) | OL MA-CS 550 mg/Day (N=1)
Accident at home (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DB MA-CS 550 mg/Day (N=2) | DB MA-CS 300 mg/Day (N=0) | DB Placebo (N=2) | OL MA-CS 550 mg/Day (N=1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other